CLINICAL TRIAL: NCT00651300
Title: A Multicentre, Double-Blind, Placebo-Controlled Study of the Recovery Benefits Following Treatment With a Cox-2 Regimen in Patients Undergoing Elective Laparoscopic Intra-Peritoneal Abdominal Surgery
Brief Title: A Study of the Recovery Benefits After Treatment With Parecoxib/Valdecoxib in Patients Undergoing Abdominal Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description field.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PARA-0505-086; A3481026
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — parecoxib; valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Parecoxib/Valdecoxib
- Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parecoxib/Valdecoxib — A single 40mg dose of intravenous (IV) parecoxib sodium administered on Day 1 immediately before the surgical procedure as part of the Investigator's usual analgesic management practice, followed by oral doses of valdecoxib 40 mg (2 x 20 mg tablets) at 6-8 hours post-surgery on Day 1 and in the morning of Day 2 and Day 3
  Arms: Group 1
Drug: Placebo — A single dose of IV saline (placebo) administered on Day 1 immediately before the surgical procedure as part of the Investigator's usual analgesic management practice, followed by oral doses of placebo (2 x matching valdecoxib 20 mg tablets) at 6-8 hours post-surgery on Day 1 and in the morning of Day 2 and Day 3
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate morphine intake in the first 4 hours after abdominal surgery. Morphine intake is compared between patients on placebo and patients on parecoxib/valdecoxib.

DETAILED DESCRIPTION:
This study was prematurely terminated because subject recruitment was slower than expected, it was determined that the study was not going to achieve the statistical power necessary to address the primary objective. Letters were sent to the sites informing them of study termination on 26 February 2004. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years weighing at least 50 kg but no more than 110 kg undergoing elective intra-peritoneal laparoscopic abdominal surgery
* American Society of Anaesthesiologists (ASA) Physical Status I-III

Exclusion Criteria:

* Significant chronic disease, such as renal, hepatic, cardiovascular, or respiratory, which would contraindicate participation in the study or interfere with interpretation of study results
* Active gastrointestinal disease, chronic or acute renal or hepatic disorder, or known coagulation defect

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2003-04; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Total intake of morphine in first 4 hours post-surgery upon waking of patients receiving parecoxib versus control group. | 4 hours

SECONDARY OUTCOMES:
Evaluation of unplanned hospital admissions on Day 4. | 4 days
Health Outcomes Recovery Questionnaire on Days 2, 3, and 4. | 4 days
Collection of adverse events immediately before surgery, 1 and 6 hours after surgery, and on Days 2, 3, and 4. | 4 days
Length of stay on Day 1. | 1 day
Patient Satisfaction Questionnaire on Days 1 and 4. | 4 days
Quality of Recovery Score on Days 1, 2, and 3. | 3 days
Numerical Rating Scale on Days 1 (hourly for 6 hours), 2, 3, and 4. | 4 days
Modified Brief Pain Inventory on Days 2, 3, and 4. | 4 days
Readiness for discharge on Day 1. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Australia (8):
  - Pfizer Investigational Site, Port Macquarie, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Coopers Plain, Queensland
  - Pfizer Investigational Site, Townsville, Queensland
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Perth, Western Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PARA-0505-086&StudyName=A%20study%20of%20the%20recovery%20benefits%20after%20treatment%20with%20parecoxib/valdecoxib%20in%20patients%20undergoing%20abdominal%20surgery